CLINICAL TRIAL: NCT01452256
Title: Desflurane and Its Effect on Postoperative Morbidity and Mortality in Patients Undergoing Thoracic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other); Kantonsspital Münsterlingen (Other); University Hospital, Basel, Switzerland (Other); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEK-ZH Nr.2011-0092
Record Dates: First submitted 2011-08-18; First posted 2011-10-14 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Thoracic Surgery
MeSH Terms: interventions — Desflurane; Propofol

ARMS (2):
- Desflurane (Experimental): Desflurane for pharmacological conditioning
  Interventions: Drug: Desflurane
- Propofol (Experimental)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Desflurane — 4-6 Vol %
  Arms: Desflurane
Drug: Propofol — TIVA to achieve BIS value of 40-60
  Arms: Propofol

SUMMARY:
Desflurane and its effect on postoperative morbidity and mortality in patients undergoing thoracic surgery.

Halothane, enflurane, isoflurane, sevoflurane, and desflurane are volatile anesthetics, a group of general anesthetics. Because of the hypnotic effects of these agents, attention has mainly focused on the central nervous system. In the last 10 years, however, numerous studies have reported that volatile anesthetic agents interact with membrane structures of the myocardium and thereby attenuate cardiac mechanical dysfunction and limit ultrastructural abnormality on reperfusion after prolonged ischemia in the myocyte. Anesthetic-induced preconditioning has become a main topic in cardiac research worldwide

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: • Elective thoracic surgery (thoracotomy, thoracoscopy)

* Lung resection
* One-lung ventilation
* Adults (18-80 years of age)
* ASA classification I - III
* Written consent (signature from patient)

Exclusion criteria:

* Known hypersensitivity or suspected allergy to propofol, soja or egg proteins
* Known hypersensitivity to volatile anesthetics (malignant hyperthermia)
* Medication with high dosage of statins
* Therapy with cyclosporin
* Severe renal impairment (GFR < 30 ml/min)
* Oral steroid treatment at present or stopped less than 3 months before surgery
* Inflammatory processes (non-pulmonary or pulmonary): elevated C-reactive protein level (> 20 mg/l) or leukocytosis (leukocytes > 10x103/?l) or body temperature > 37°C)
* Pregnancy
* Breast feeding
* The subject must not be involved in any other clinical trial during the course of this trial, nor within a period of 30 days prior to its beginning or 30 days after its completion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Major complications as defined as ≥ grade IIIa according to classification of surgical complications from Dindo et al. after lung resection with one-lung ventilation during hospitalization | postoperative phase until discharge; 6 month after surgery

SECONDARY OUTCOMES:
Major complications ≥ grade IIIa according to classification of surgical complications from Dindo et al. after dimissio up to 6 months after surgery | postoperative phase until discharge, 6 month postoperative
Perioperative inflammatory mediators TNF-α, IL-6, IL-8, sICAM-1, MCP-1, MIP-2 in blood (correlation to complications ≥ grade IIIa according to classification of surgical complications from Dindo et al. during hospitalization) | postoperative phase until discharge

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Beatrice Beck Schimmer, Professor, Principal Investigator — University Hospital Zurich, Division of Anaesthesiology
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Neff TA, Braun J, Rana D, Puhan M, Filipovic M, Seeberger M, Stuber F, Neff SB, Beck-Schimmer B, Schlapfer M. Interleukin-6 Is an Early Plasma Marker of Severe Postoperative Complications in Thoracic Surgery: Exploratory Results From a Substudy of a Randomized Controlled Multicenter Trial. Anesth Analg. 2022 Jan 1;134(1):123-132. doi: 10.1213/ANE.0000000000005639. PMID 34132704